CLINICAL TRIAL: NCT03649061
Title: Effectiveness of a Combination of Methotrexate and a Step Down Glucocorticoid Regimen (COBRA-Slim) for Remission Induction in Patients With Early Rheumatoid Arthritis (RA), With or Without Fast Access to 24 Weeks of Tumor Necrosis Factor (TNF) Blockade in Insufficient Responders, a Randomized, Multicenter, Pragmatic Trial
Brief Title: COBRA-Slim With or Without Fast Access to TNF Blockade for Remission Induction in Early RA
Acronym: CareRA2020
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: P. Verschueren (Other)
Collaborators: Belgium Health Care Knowledge Centre (Other Government)
Responsible Party: Sponsor-Investigator, P. Verschueren, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCE-16002; 2017-004054-41 (EudraCT Number)
Record Dates: First submitted 2018-07-30; First posted 2018-08-28 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Arthritis, Rheumatoid
Keywords: COBRA-Slim; Accelerated access to anti-TNF; treat to target; remission induction
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Intervention Model Description: Insufficient responders to a COBRA-Slim strategy, defined as not reaching low disease activity based on DAS28 CRP from week 8 until week 32 or not reaching remission based on DAS28 CRP at week 32, will be randomly assigned to one of the two arms.
  Randomization will be balanced according to time-point of randomization, baseline (BL) disease activity and Anti-Citrullinated Protein Antibody (ACPA) and Rheumatoid Factor (RF) status to ensure comparability of the treatment groups with respect to these prognostic variables.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard COBRA-Slim induction (Active Comparator): Leflunomide 10mg PO daily added to the COBRA-Slim scheme (Methotrexate 15 mg PO weekly, Step down scheme of GC: 30-20-12,5-10-7,5-5 mg prednisone PO daily, each for 7 days except for the lowest dose of 5 mg, this will be maintained until w28 and then tapered to 2.5 mg daily for two weeks before stopping completely.)
  Interventions: Drug: Leflunomide 10 milligram (MG)
- COBRA-Slim Bio-induction (Experimental): Etanercept 50mg subcutaneous (SC) weekly added for 24 weeks to COBRA-Slim scheme (Methotrexate 15 mg PO weekly, Step down scheme of GC: 30-20-12,5-10-7,5-5 mg prednisone PO daily, each for 7 days except for the lowest dose of 5 mg, this will be maintained until w28 and then tapered to 2.5 mg daily for two weeks before stopping completely.)
  Interventions: Drug: Etanercept 50 MG/ML

INTERVENTIONS:
Drug: Etanercept 50 MG/ML — Etanercept 50mg subcutaneous (SC) weekly added for 24 weeks to COBRA-Slim scheme
  Arms: COBRA-Slim Bio-induction
Drug: Leflunomide 10 milligram (MG) — Leflunomide 10mg PO daily added to the COBRA-Slim scheme
  Arms: standard COBRA-Slim induction

SUMMARY:
In the Care in Rheumatoid Arthritis (CareRA) trial (NCT01172639) about 70% of early RA patients are in remission at the 2 year evaluation point independent of the combination scheme used.

Interesting to see is that the 30% of insufficient responders can be identified in an early stage of the treatment course.

The purpose of the present study is to investigate if, for patients with an insufficient response to a COBRA-Slim regimen, accelerated access to a short course of anti-TNF therapy already early after treatment initiation (from w8 until w32) could improve outcomes compared to a more traditional treat to target sequence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of RA as defined by the American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) 2010 criteria for early RA
* Early RA defined by a diagnosis made ≤ 1 year ago.
* Use a reliable method of contraception for women of childbearing potential to be evaluated as in daily clinical practice
* Able and willing to give written informed consent and to participate in the study
* Understanding and able to write Dutch or French

Exclusion Criteria:

* Previous treatment with:

  * Methotrexate (MTX) or leflunomide
  * cyclophosphamide, azathioprine or cyclosporine
  * sulphasalazine (SSZ) for more than 3 weeks
  * hydroxychloroquine for more than 6 weeks
  * oral Glucocorticoids (GC) for more than 4 weeks within 4 months before screening
  * oral GC at a daily dosage of more than 10 mg prednisone equivalent within 4 weeks before baseline
  * oral GC at a daily dosage equal to or less than 10 mg prednisone equivalent within 2 weeks before baseline
  * intra-articular GC within 4 weeks before BL
  * an investigational drug for the treatment/prevention of RA
* History of chronic heart failure
* History of severe infections or chronic infection
* History of malignant neoplasm within 5 years
* Contra indications for GC
* Contra indications for TNF blocking agents
* Contra indications for MTX or leflunomide
* Psoriatic Arthritis
* Underlying cardiac, pulmonary, metabolic, renal or gastrointestinal conditions, chronic or latent infectious diseases or immune deficiency which in the opinion of the investigator places the patient at an unacceptable risk for participation in the study
* Pregnancy, breastfeeding or no use of a reliable method of contraception for woman of childbearing potential (as in daily clinical practice)
* Alcohol or drug abuse
* Active tuberculosis (TB)
* Latent TB unless adequate prophylactic treatment is given according to local guidelines
* No access to the Belgian Health Insurance system-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Verschueren, MD, PhD, Principal Investigator — UZ Leuven
Locations (19):
- Belgium (19):
  - Imelda Ziekenhuis Bonheiden, Bonheiden, Antwerpen
  - AZ Herentals, Herentals, Antwerpen
  - ZNA Jan Palfijn, Merksem, Antwerpen
  - GHdC Saint Joseph, Gilly, Henegouwen
  - Reuma centrum Genk, Genk, Limburg
  - Reuma Clinic Genk, Genk, Limburg
  - Reuma Instituut Hasselt, Hasselt, Limburg
  - CHU UCL Namur ASBL Site Godinne, Yvoir, Namur
  - OLV Ziekenhuis Aalst, Aalst, Oost Vlaanderen
  - Regionaal Ziekenhuis Heilig Hart Leuven, Leuven, Vlaams Brabant
  - UZ Leuven, Leuven, Vlaams Brabant
  - AZ Jan Portaels, Vilvoorde, Vlaams Brabant
  - AZ St Lucas Brugge, Bruges, West Vlaanderen
  - AZ Sint Jan Brugge, Bruges, West-Vlaanderen
  - CHU Saint Pierre, Brussels
  - Cliniques Universitaire Saint Luc (UCL), Brussels
  - Hôpital Erasme-ULB, Brussels
  - UZ Brussel, Brussels
  - CHU Liège, Liège

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van der Elst K, De Cock D, Vecoven E, Arat S, Meyfroidt S, Joly J, Moons P, Verschueren P, Westhovens R, CareRA Study Group. Are illness perception and coping style associated with the delay between symptom onset and the first general practitioner consultation in early rheumatoid arthritis management? An exploratory study within the CareRA trial. Scand J Rheumatol. 2016;45(3):171-8. doi: 10.3109/03009742.2015.1074278. Epub 2015 Sep 23. PMID 26399601
- [Background] Verschueren P, Esselens G, Westhovens R. Predictors of remission, normalized physical function, and changes in the working situation during follow-up of patients with early rheumatoid arthritis: an observational study. Scand J Rheumatol. 2009 May-Jun;38(3):166-72. doi: 10.1080/03009740802484846. PMID 19169906
- [Result] Verschueren P, Westhovens R. The use of glucocorticoids in early rheumatoid arthritis. Rheumatology (Oxford). 2018 Aug 1;57(8):1316-1317. doi: 10.1093/rheumatology/kex271. No abstract available. PMID 28968687
- [Result] Verschueren P, De Cock D, Corluy L, Joos R, Langenaken C, Taelman V, Raeman F, Ravelingien I, Vandevyvere K, Lenaerts J, Geens E, Geusens P, Vanhoof J, Durnez A, Remans J, Vander Cruyssen B, Van Essche E, Sileghem A, De Brabanter G, Joly J, Meyfroidt S, Van der Elst K, Westhovens R. Effectiveness of methotrexate with step-down glucocorticoid remission induction (COBRA Slim) versus other intensive treatment strategies for early rheumatoid arthritis in a treat-to-target approach: 1-year results of CareRA, a randomised pragmatic open-label superiority trial. Ann Rheum Dis. 2017 Mar;76(3):511-520. doi: 10.1136/annrheumdis-2016-209212. Epub 2016 Jul 18. PMID 27432356
- [Result] De Cock D, Van der Elst K, Meyfroidt S, Verschueren P, Westhovens R. The optimal combination therapy for the treatment of early rheumatoid arthritis. Expert Opin Pharmacother. 2015;16(11):1615-25. doi: 10.1517/14656566.2015.1056735. Epub 2015 Jun 10. PMID 26058860
- [Result] Verschueren P, De Cock D, Corluy L, Joos R, Langenaken C, Taelman V, Raeman F, Ravelingien I, Vandevyvere K, Lenaerts J, Geens E, Geusens P, Vanhoof J, Durnez A, Remans J, Vander Cruyssen B, Van Essche E, Sileghem A, De Brabanter G, Joly J, Van der Elst K, Meyfroidt S, Westhovens R; CareRA study group. Patients lacking classical poor prognostic markers might also benefit from a step-down glucocorticoid bridging scheme in early rheumatoid arthritis: week 16 results from the randomized multicenter CareRA trial. Arthritis Res Ther. 2015 Apr 9;17(1):97. doi: 10.1186/s13075-015-0611-8. PMID 25889222
- [Result] Meyfroidt S, Van der Elst K, De Cock D, Joly J, Westhovens R, Hulscher M, Verschueren P. Patient experiences with intensive combination-treatment strategies with glucocorticoids for early rheumatoid arthritis. Patient Educ Couns. 2015 Mar;98(3):384-90. doi: 10.1016/j.pec.2014.11.011. Epub 2014 Nov 20. PMID 25483574
- [Result] Verschueren P, De Cock D, Corluy L, Joos R, Langenaken C, Taelman V, Raeman F, Ravelingien I, Vandevyvere K, Lenaerts J, Geens E, Geusens P, Vanhoof J, Durnez A, Remans J, Vander Cruyssen B, Van Essche E, Sileghem A, De Brabanter G, Joly J, Meyfroidt S, Van der Elst K, Westhovens R. Methotrexate in combination with other DMARDs is not superior to methotrexate alone for remission induction with moderate-to-high-dose glucocorticoid bridging in early rheumatoid arthritis after 16 weeks of treatment: the CareRA trial. Ann Rheum Dis. 2015 Jan;74(1):27-34. doi: 10.1136/annrheumdis-2014-205489. Epub 2014 Oct 30. PMID 25359382
- [Result] Meyfroidt S, van Hulst L, De Cock D, Van der Elst K, Joly J, Westhovens R, Hulscher M, Verschueren P. Factors influencing the prescription of intensive combination treatment strategies for early rheumatoid arthritis. Scand J Rheumatol. 2014;43(4):265-72. doi: 10.3109/03009742.2013.863382. Epub 2014 Feb 24. PMID 24559216
- [Result] Westhovens R, Verschueren P. Rheumatoid arthritis: defining remission in patients with RA in clinical practice. Nat Rev Rheumatol. 2012 Aug;8(8):445-7. doi: 10.1038/nrrheum.2012.111. Epub 2012 Jul 3. No abstract available. PMID 22751567
- [Result] Verschueren P, Westhovens R. Optimal care for early RA patients: the challenge of translating scientific data into clinical practice. Rheumatology (Oxford). 2011 Jul;50(7):1194-200. doi: 10.1093/rheumatology/ker131. Epub 2011 Mar 30. PMID 21454307
- [Result] Durez P, Malghem J, Nzeusseu Toukap A, Depresseux G, Lauwerys BR, Westhovens R, Luyten FP, Corluy L, Houssiau FA, Verschueren P. Treatment of early rheumatoid arthritis: a randomized magnetic resonance imaging study comparing the effects of methotrexate alone, methotrexate in combination with infliximab, and methotrexate in combination with intravenous pulse methylprednisolone. Arthritis Rheum. 2007 Dec;56(12):3919-27. doi: 10.1002/art.23055. PMID 18050189
- [Result] Boers M, Verhoeven AC, Markusse HM, van de Laar MA, Westhovens R, van Denderen JC, van Zeben D, Dijkmans BA, Peeters AJ, Jacobs P, van den Brink HR, Schouten HJ, van der Heijde DM, Boonen A, van der Linden S. Randomised comparison of combined step-down prednisolone, methotrexate and sulphasalazine with sulphasalazine alone in early rheumatoid arthritis. Lancet. 1997 Aug 2;350(9074):309-18. doi: 10.1016/S0140-6736(97)01300-7. PMID 9251634
- [Derived] Bertrand D, Joly J, Neerinckx B, Durez P, Lenaerts J, Joos R, Thevissen K, Zwaenepoel T, Vanhoof J, Di Romana S, Taelman V, Van Essche E, Corluy L, Ribbens C, Vanden Berghe M, Devinck M, Ajeganova S, Durnez A, Boutsen Y, Margaux J, Peene I, Van Offel J, Doumen M, Pazmino S, De Meyst E, Kulyk M, Creten N, Westhovens R, Verschueren P; CareRA2020 Study group. Effectiveness of methotrexate and bridging glucocorticoids with or without early introduction of a 6-month course of etanercept in early RA: results of the 2-year, pragmatic, randomised CareRA2020 trial. RMD Open. 2024 Aug 7;10(3):e004535. doi: 10.1136/rmdopen-2024-004535. PMID 39117445

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 284 patients screened, 276 were eligible for the trial and 122 met the criteria of early insufficient responders to an initial COBRA-Slim remission induction regimen. Of this last group 112 patients were randomized, however 2 were considered randomization errors, 10 patients were eligible for randomization but were not randomized per investigator decision.
Pre-assignment Details: All patients received a COBRA-Slim remission induction regimen, consisting of methotrexate (MTX) with a step-down scheme of glucocorticosteroids (GC).
  Patient not reaching low disease activity, based on DAS28CRP, before week 32 or DAS28CRP remission at week 32 were considered early insufficient responders and were eligible for randomization.
Period: Overall Study
Arm/Group | Standard COBRA-Slim Induction | COBRA-Slim Bio-induction
Started | 55 | 55
Completed | 46 | 46
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard COBRA-Slim Induction | COBRA-Slim Bio-induction | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 48 | 91
  >=65 years | 12 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (13.1) | 52.5 (12.9) | 52.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 79
  Male | 14 | 17 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 55 | 55 | 110
smoking [Count of Participants; unit: Participants]
  never | 22 | 19 | 41
  past | 14 | 13 | 27
  current | 19 | 23 | 42
Rheumatoid factor (RF)/Anti-citrullinated protein antibodies (ACPA ) status [Count of Participants; unit: Participants]
  positive | 42 | 41 | 83
  negative | 13 | 14 | 27
Disease activity (DAS28CRP) [Mean (Standard Deviation); unit: units on a scale] — Disease activity score based on a 28 joint count (Tender and Swollen joints) and C-Reactive Proteine (CRP) value.
  Scale range 0.0 to 9.4.
  Scale interpretation:
  * Remission: value below 2.6
  * Low disease activity: from 2.6 till 3.2 (included)
  * Moderate disease activity: above 3.2 till 5.1
  * High disease activity: above 5.1
  units on a scale | 5.4 (1.1) | 5.2 (1.3) | 5.3 (1.2)
Disease duration [Median (Inter-Quartile Range); unit: days] | 7.0 [2.5 to 20.0] | 7.0 [2.5 to 19.5] | 7.0 [2.3 to 19.8]

OUTCOME MEASURES:

1. Primary Outcome: Area Under Curve (AUC) of Disease Activity Score Based on a 28 Jointcount and C-reactive Protein (DAS28CRP)
Description: Analysis was based on an intention to treat population, which focused on all patients randomized into the study, irrespective if they actually received the randomized treatment. Fifty-five patients were allocated to Standard COBRA-Slim and 55 to COBRA-Slim Bio-induction.
  This measure is an indication of the total disease-activity over time or long-term effectiveness, a higher area under the curve indicates a higher disease activity over time and so a lower effectiveness over the time frame of the trial.
  The scale range for the duration of the trial (104 weeks) is 0.0 to 977.6
  * remission: value below 270.4
  * low disease activity: from 270.4 till 332.8 (included)
  * moderate disease activity: above 332.8 till 530.4
  * high disease activity: above 530.4
Time Frame: baseline, w4, w8, w16, w24, w32, w40, w52, w64, w78, w92 and w104
Population: intention to treat (ITT) population
Measure: Mean (95% Confidence Interval); unit: units on a scale*week
Arm/Group | Standard COBRA-Slim Induction | COBRA-Slim Bio-induction
Number analyzed (Participants) | 55 | 55
units on a scale*week | 297.4 [277.1 to 317.7] | 300.7 [282.3 to 319.1]
Statistical Analysis 1: Comparison: Standard COBRA-Slim Induction vs COBRA-Slim Bio-induction; To compare the two randomization groups, a linear mixed model with DAS28-CRP as outcome (Bell et al. 2014), including random intercepts per patient, adjusted for baseline DAS28-CRP, randomization timepoint, and RF and/or ACPA seropositivity was used; Test type: Superiority; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Proportion of Insufficient Responders Achieving Remission (DAS28CRP<2.6) 28 Weeks After Randomization (Short Term Efficacy) to Either COBRA-Slim Bio-Induction or Standard COBRA-Slim Induction
Description: Short-time efficacy of disease activity based on a swollen and tender joint count of 28 joints and C-reactive proteine (scale range 0.0 to 9.4; remission: value below 2.6; low disease activity: from 2.6 till 3.2 (included); moderate disease activity: above 3.2 till 5.1; high disease activity: above 5.1).
Time Frame: From randomization till 28 weeks after randomization.
Population: intention to treat (ITT) population
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Standard COBRA-Slim Induction | COBRA-Slim Bio-induction
Number analyzed (Participants) | 55 | 55
participants | 24 [17 to 32] | 32 [24 to 40]
Statistical Analysis 1: Comparison: Standard COBRA-Slim Induction vs COBRA-Slim Bio-induction; A binomial generalized linear mixed effect model for repeated measures of remission from randomization up until 28 weeks after was carried out, with adjustment for baseline DAS28-CRP, moment of randomization, and RF and/or ACPA seropositivity; Test type: Superiority; p < 0.05, Mixed Models Analysis

3. Secondary Outcome: Proportion of Patients in Remission Defined as DAS28CRP<2.6
Description: as for outcome 2
Time Frame: at week 104
Population: intention to treat (ITT) population
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Standard COBRA-Slim Induction | COBRA-Slim Bio-induction
Number analyzed (Participants) | 55 | 55
participants | 38 [30 to 44] | 30 [22 to 37]

4. Secondary Outcome: Proportion of Patients Achieving a EULAR Response
Description: proportion of patients achieving a EULAR response, based on actual disease activity on a tender/swollen joint count and C-reactive proteine (DAS28-CRP) 28 weeks after randomization and improvement in DAS28-CRP from baseline.
  The EULAR response criteria classify patients as good, moderate or non-responders, using the individual amount of change in the DAS28-CRP and the DAS28-CRP value (low, moderate, or high) reached according to the following tabel:
  DAS28-CRP at endpoint improvement in DAS28-CRP from baseline <=1,2 >0,6 and <= 1,2 <=0,6 <= 3,2 good moderate none >3,2 and <= 5,1 moderate moderate none >5,1 moderate none none Additionally all patients with a good response were also included in the number of participants with at least a moderate response.
Time Frame: at 28 weeks after randomization
Population: Intention to treat (ITT) population
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Standard COBRA-Slim Induction | COBRA-Slim Bio-induction
Number analyzed (Participants) | 55 | 55
participants
  Good Response | 26 [18 to 34] | 25 [18 to 33]
  Moderate Response | 41 [32 to 47] | 40 [32 to 46]

5. Secondary Outcome: Proportion of Patients Achieving a EULAR Response
Description: proportion of patients achieving a EULAR response, based on actual disease activity on a tender/swollen joint count and C-reactive proteine (DAS28-CRP) at week 104 and improvement in DAS28-CRP from baseline.
  The EULAR response criteria classify patients as good, moderate or non-responders, using the individual amount of change in the DAS28-CRP and the DAS28-CRP value (low, moderate, or high) reached according to the following tabel:
  DAS28-CRP at endpoint improvement in DAS28-CRP from baseline <=1,2 >0,6 and <= 1,2 <=0,6 <= 3,2 good moderate none >3,2 and <= 5,1 moderate moderate none >5,1 moderate none none Additionally all patients with a good response were also included in the number of participants with at least a moderate response.
Time Frame: at week 104
Population: Intention to treat (ITT) population
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Standard COBRA-Slim Induction | COBRA-Slim Bio-induction
Number analyzed (Participants) | 55 | 55
participants
  Good Response | 42 [35 to 48] | 34 [26 to 41]
  Moderate Response | 52 [45 to 54] | 49 [42 to 52]

6. Secondary Outcome: Health Assessment Questionnaire (HAQ) Response
Description: HAQ measures physical function as reported by the patient, total score range from 0-3 of which higher scores represent worse physical function.
Time Frame: at 28 weeks after randomization
Population: Intention to treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard COBRA-Slim Induction | COBRA-Slim Bio-induction
Number analyzed (Participants) | 55 | 55
score on a scale | 0.7 (0.7) | 0.8 (0.7)

7. Secondary Outcome: Health Assessment Questionnaire (HAQ) Response
Description: as for outcome 6
Time Frame: at week 104
Population: Intention to treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard COBRA-Slim Induction | COBRA-Slim Bio-induction
Number analyzed (Participants) | 55 | 55
score on a scale | 0.7 (0.7) | 0.9 (0.7)

8. Secondary Outcome: Radiographic Progression
Description: Radiographic progression at week 52 is scored according to the Sharp-Van der Heijde score (SvdH).
  The SvdH method scores the presence of erosions in 16 joints of hands and wrists (graded from 0 to 5), and in 6 joints of the feet (graded from 0 to 10), and the presence of joint space narrowing in 15 joints of the hands and wrists (graded from 0 to 4) and in 6 joints of the feet (graded from 0 to 4). The maximal range is 280 units for erosion and 168 units for joint space narrowing, summing up to 448 units for the total score.
  The progression is calculated by subtracting the total score at week 52 minus the total score at baseline (ranging from 0 to 448) Higher values in each (sub) scale represents a worse outcome.
Time Frame: at week 52
Population: Intention to treat (ITT) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard COBRA-Slim Induction | COBRA-Slim Bio-induction
Number analyzed (Participants) | 55 | 55
units on a scale | 0.5 (1.2) | 0.3 (0.9)

9. Secondary Outcome: Radiographic Progression
Description: Radiographic progression at week 104 is scored according to the Sharp-Van der Heijde score (SvdH).
  The SvdH method scores the presence of erosions in 16 joints of hands and wrists (graded from 0 to 5), and in 6 joints of the feet (graded from 0 to 10), and the presence of joint space narrowing in 15 joints of the hands and wrists (graded from 0 to 4) and in 6 joints of the feet (graded from 0 to 4). The maximal range is 280 units for erosion and 168 units for joint space narrowing, summing up to 448 units for the total score.
  The progression is calculated by subtracting the total score at week 104 minus the total score at baseline (ranging from 0 to 448) Higher values in each (sub) scale represents a worse outcome.
Time Frame: at week 104
Population: Intention to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard COBRA-Slim Induction | COBRA-Slim Bio-induction
Number analyzed (Participants) | 55 | 55
units on a scale | 0.7 (2.1) | 0.8 (1.7)

ADVERSE EVENTS:
Time Frame: (Serious) adverse reactions or events of interest are collected over the duration of the trial e.g. 2 years (from screening till w104)
Description: In the CareRA2020 trial, only (serious) events related to rheumatoid arthritis (RA), the RA treatment, or in case of an event of special interest (as specified in the protocol and including deaths) are to be reported according to the protocol. Collection of these reactions was done by delegated study staff questioning the patient at each visit.
Arm/Group | Standard COBRA-Slim Induction | COBRA-Slim Bio-induction
All-Cause Mortality (participants affected / at risk) | 1/55 | 1/55
Serious Adverse Events (participants affected / at risk) | 4/55 | 5/55
Other Adverse Events (participants affected / at risk) | 43/55 | 47/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard COBRA-Slim Induction (N=55) | COBRA-Slim Bio-induction (N=55)
aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
cerobrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
psychiatric decompensation (Psychiatric disorders) | 0 (0) | 1 (1)
bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard COBRA-Slim Induction (N=55) | COBRA-Slim Bio-induction (N=55)
fatigue (General disorders) | 12 (12) | 13 (13)
injection site erythema (General disorders) | 1 (1) | 3 (3)
pyrexia (General disorders) | 0 (0) | 4 (5)
palpitations (Cardiac disorders) | 0 (0) | 4 (4)
headache (Nervous system disorders) | 1 (1) | 3 (4)
nausea (Gastrointestinal disorders) | 8 (11) | 14 (17)
abdominal discomfort (Gastrointestinal disorders) | 5 (5) | 6 (6)
diarrhoea (Gastrointestinal disorders) | 10 (11) | 6 (7)
abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 4 (5)
gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2)
hepatic function abnormal (Hepatobiliary disorders) | 14 (18) | 9 (12)
alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
acne (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2)
nasopharyngitis (Infections and infestations) | 4 (4) | 3 (4)
COVID-19 (Infections and infestations) | 2 (2) | 6 (6)
bronchitis (Infections and infestations) | 3 (4) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/PI may only publish the Results provided that Sponsor has duly published the main Study publication. Once the main Study publication has been duly published by the Sponsor, Institution/PI are entitled to publish the Results provided that Sponsor has granted its prior written approval with Institution's/PI's proposed publication. If SPONSOR did not respond within 90 days, the institution/PI may proceed with the publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT03649061/Prot_SAP_000.pdf